CLINICAL TRIAL: NCT01227525
Title: Assessing Pain Behaviors of Children Receiving Local Anesthesia Using VibraJect Attachment
Brief Title: Assessing the Benefits of the Vibraject Attachment
Acronym: Vibraject
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keith Allen, PhD (Other)
Responsible Party: Sponsor-Investigator, Keith Allen, PhD, Secondary Investigator, University of Nebraska
Organization: University of Nebraska (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 535-07-FB
Record Dates: First submitted 2009-04-27; First posted 2010-10-25 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vibraject — The VibraJect clips onto the barrel of a conventional and intraligamentary dental syringe (and some disposable syringes) and vibrates the needle at a high frequency while injections are administered.

SUMMARY:
Behavioral and physiologic observations suggest that the injection of local anesthetic is among the most feared or anxiety producing procedures during dental intervention. Discomfort during the injection is currently reduced by pharmacologic or mechanical methods. No technique has proven to be effective for every patient. The VibraJect LLC (USA) was first introduced in 1995 and was developed under the hypothesis that a vibrating needle would stimulate large diameter nerve fibers and thereby close the gate to smaller nerves carrying the pain signal from the injection site. Studies on adult patients have been promising. The purpose of this study is to investigate the efficacy of the VibraJect dental syringe attachment in reducing injection discomfort and procedural anxiety in the pediatric dental population.

DETAILED DESCRIPTION:
One hundred children will be recruited from the UNMC Pediatric Dentistry clinic. Eligible children will be selected from the 4-6 year group who are scheduled for routine dental restorative treatment and who have or have never received a dental injection. Each patient will randomly participate in either a control or experimental condition. The device will be attached for both conditions. During the control injection, the dentist will perform the dental injection as usual. During the experimental injection, the dentist will activate the attached device and perform the injection. Immediately following each injection, the patient will rate the pain on a visual analog scale and a trained observer will rate the child's behavior on a Frankl behavior scale. A videotape of the procedure will be reviewed by an independent dentist who will evaluate the child's response and any perceived disruptive behavior. This observer will be blind to whether the instrument is functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Attending the UNMC pediatric dentistry clinic for dental restorations requiring injection of local anesthetic for restorative procedures with or without use of inhalation anesthesia but without physical restraint
2. age 4 to 8

Exclusion Criteria:

1. No parent or legal guardian is present
2. Parent does not give consent
3. Non-English speaking participants will be excluded because PI is English speaking and this study needs behavior guidance of children that only the dentist can deliver and not an interpreter.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Observed disruptive behavior | 1 Year

SECONDARY OUTCOMES:
Behavior ratings by dentist of cooperative behavior | 1 Year
subjective pain ratings on visual analogue scale | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Brandi Roeber, DDS, Principal Investigator — University of Nebraska